CLINICAL TRIAL: NCT04779203
Title: Prospective Study Comparing Standard Extraction Drilling With Osseodensification for Dental Implant Placement
Brief Title: Study Comparing Osseodensification With Standard Drilling
Acronym: OD/SD
Status: Completed | Type: Observational
Sponsor: Jackson Implant Surgery (Industry)
Responsible Party: Principal Investigator, Salah Huwais, Principal Investigator, Jackson Implant Surgery
Other Study IDs: JacksonImplantS
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Tooth Loss
Keywords: Osseodensification, Standard Extraction Drilling; Implant Primary stability, Implant Secondary Stability
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Osseodensification: Osseodensification is a novel, biomechanical osteotomy preparation technique that preserves bone through a non-excavating drilling process utilizing specially designed burs with a tapered geometry and specially designed flutes progressively expand the osteotomy whilst compacting bone into its walls and apex.
  Interventions: Device: Osseodensification Densah Bur
- Standard Drilling: Utilizing conventional drilling technique with standard bone drilling techniques.
  Interventions: Device: Osseodensification Densah Bur

INTERVENTIONS:
Device: Osseodensification Densah Bur — Implants placed with osseodensification surgical drilling compared to those placed with subtractive conventional drilling technique in a split-mouth design will result: 1) in the same insertion torque values and; 2) in the same implant stability quotient values when measured immediately after implant placement and after 1, 2, 3, 4, 5, 6, 7, 8, and 12 weeks.
  Other Names: Densah Bur

SUMMARY:
The purpose of this study is to examine how Osseodensification, a well-defined bone preparation procedure utilizing special densifying burs (a tool to prepare bone) compares to the standard drilling procedure utilizing regular bone drills, to possibly enhance dental implant healing.

DETAILED DESCRIPTION:
Our postulated null hypotheses is that implants placed with osseodensification surgical drilling compared to those placed with subtractive conventional drilling technique in a split-mouth design will result: 1) in the same insertion torque values and; 2) in the same implant stability quotient values when measured immediately after implant placement and after 1, 2, 3, 4, 5, 6, 7, 8, and 12 weeks.

Study Objectives:

A.Perform a prospective clinical study to investigate implant primary stability through measuring insertion torque values (IT) and Implant stability quotient (ISQ) when implants are placed using a standard drilling protocol (subtractive surgical drilling, as recommended by implant manufacturers) compared to osseodensification drilling protocol in a split-mouth design.

B.Implant stability quotient will be measured once the implant is placed (immediate), and at 1, 2, 3, 4, 5, 6, 7, 8, and 12 weeks.

C.To investigate, and analyze these two surgical drilling protocols as function of different implant manufacturers with variations in diameter and length.

D.To further track trends in the use of osseodensification surgical drilling once the patient receives the prosthodontic reconstruction.

E.To share the knowledge generated from this prospective analysis through scientific publications.

Patient selection will focus on the need of implant placement on the right and left equivalent sides of the maxilla/mandible where one side/site will receive implant(s) placed post osseodensification surgical drilling recommended by Densifying reference guide of the Densah Burs manufacturer, and the other side/site will receive implant(s) placed by the control technique, which is subtractive conventional drilling recommended by the specific implant manufacturer.

Written consent will be provided, explained and signed by participating patients.

After Dental Implant procedure, participating patients will be asked to participate in 6-12 weekly follow visits.

Subjects Selection and Study Procedures:

Study will include 23 patients. Patients should not be in another research study or have not been in any other research study in the last 90 days. They cannot be in this study if they are abusing any drugs.

Patient selection will focus on the need of implant placement on the right and left equivalent sides of the maxilla/ mandible where one side/site will receive implant(s) placed by osseodensification surgical drilling, and the other side/site will receive implant(s) placed by the control surgical technique, which is subtractive conventional drilling recommended by the implant manufacturer.

Written consent will be provided, explained and signed by participating patients.

After Dental Implant procedure, participating patients will be asked to participate in 6-12 weekly follow-up visits.

Subjects Selection and Study Procedures:

Study will include 23 patients. Patients should not be in another research study or have not been in any other research study in the last 90 days. They cannot be in this study if they are abusing any drugs.

Patient selection will focus on the need of implant placement on the right and left equivalent sides of the maxilla/mandible where one side/site will receive implant(s) placed by osseodensification surgical drilling according to the manufacturer Densifying Reference Guide, and the other side/site will receive implant(s) placed by the control surgical technique, which is subtractive conventional drilling recommended by the implant manufacturer.

Written consent will be provided, explained and signed by participating patients.

After Dental Implant procedure, participating patients will be asked to participate in 6-12 weekly follow visits.

Study Procedures:

1. The implants will both be placed in the upper or lower jaw. The type of placement preparation of the first implant will be determined by chance (like flipping a coin) with other preparation for the second implant site. Implant primary stability will be measured initially by measuring insertion torque values utilizing a commercially available and validated clinical torque indicator.
2. Implant placement procedure will follow the standard of care for both implants for pain management, aftercare and infection control.
3. During the weekly follow-up visits over 6-12 weeks, we will conduct a non-invasive measurement of Implant secondary stability utilizing the Osstell device. Osstell is a resonance frequency tester, which will create a gentle vibration in the implant and measure how much if any the implant moves with the vibration. The device will not loosen the implant. The standard of care is after confirming implant healing and high secondary stability is to initiate yearly follow up as needed.

ELIGIBILITY:
Inclusion Criteria:

* Patient needs an implant placements in both maxilla and mandible.
* Patients are medically stable.

Exclusion Criteria:

* Drug Abuse
* Patient should not have been in any other research study in the last 90 days from the study starting date.

Ages: 22 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study will include 23 patients. Patients should not be in another research study or have not been in any other research study in the last 90 days. They cannot be in this study if they are abusing any drugs.
  Patients are older than 22 years, medically Stable Patients should not be in another research study or have not been in any other research study in the last 90 days.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Implant Primary Stability | Day 0
  Implant primary stability is a mechanical parameters that reflects implant stability Day of surgery. Implant primary stability is measured by measuring implant insertion torque (measured during implant insertion with a torque wrench)
Implant Secondary Stability | 1-16 weeks
  During the weekly follow-up visits over 1-12 weeks, we will conduct a non-invasive measurement of implant secondary stability (correlated to BIC) utilizing the Osstell device. Osstell is a resonance frequency tester, which will create a gentle vibration in the implant and measure how much if any the implant moves with the vibration. The device will not loosen the implant. We will measure weekly. The standard of care is measurement of implant stability at 6-12 weeks post implant placement with yearly follow up as needed.

SECONDARY OUTCOMES:
Cumulative implant survival rate | 10-16 weeks
  Implant Osseointegration success rate
Bone Instrumentation effect on different implant geometry | 1-16 weeks
  Study, and analyze these two surgical drilling protocols as function of different implant manufacturers with variations in diameter and length.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Huwais, DDS, Principal Investigator — Jackson Implant Surgery
Locations (1):
- Salah Huwais, DDS, PLLC, Jackson, Michigan, United States

IPD SHARING:
Plan to Share IPD: No